CLINICAL TRIAL: NCT00003662
Title: A Pilot Study of Unrelated Umbilical Cord Blood Transplantation in Adults and Children With Bone Marrow Failure Syndromes or Inherited Metabolic or Hematologic Diseases
Brief Title: Umbilical Cord Blood Transplantation in Treating Patients With Hematologic Cancer or Other Hematologic or Metabolic Diseases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066755; P30CA016056 (NIH); RPCI-RP-9803; NCI-G98-1486
Record Dates: First submitted 1999-11-01; First posted 2004-08-04 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Graft Versus Host Disease; Leukemia; Myelodysplastic Syndromes; Thymic Carcinoma
Keywords: noninvasive thymoma and thymic carcinoma; recurrent thymoma and thymic carcinoma; refractory anemia; refractory anemia with ringed sideroblasts; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; graft versus host disease; childhood myelodysplastic syndromes
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Myelodysplastic Syndromes; Thymoma; Anemia, Refractory | interventions — Antilymphocyte Serum; Busulfan; Cyclophosphamide; Cyclosporine; Melphalan; Methylprednisolone; Cord Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: anti-thymocyte globulin
Drug: busulfan
Drug: cyclophosphamide
Drug: cyclosporine
Drug: melphalan
Drug: methylprednisolone
Procedure: umbilical cord blood transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Umbilical cord blood transplantation may be able to replace cells destroyed by chemotherapy or radiation therapy.

PURPOSE: Phase II trial to study the effectiveness of umbilical cord blood transplantation in treating patients who have hematologic cancer or other hematologic or metabolic diseases.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the rates of durable engraftment in patients with severe aplastic anemia, myelodysplastic syndrome, inborn errors of metabolism, or inherited hematopoietic disorders refractory to medical management, who are undergoing high dose chemoradiotherapy followed by unrelated cord blood (UCB) transplantation. II. Determine the incidence and severity of acute and chronic graft-versus-host disease in these patients. III. Monitor overall and event-free survival of these patients. IV. Evaluate rate and quality of immunologic reconstitution of these patients. V. Determine whether nucleated cell or progenitor cell content of the graft is predictive of engraftment.

OUTLINE: This is a multicenter study. Patients are stratified according to low vs high weight. Patients with severe aplastic anemia, myelodysplastic syndrome, or bone marrow failure receive cyclophosphamide IV over 1 hour on days -6 to -3 or melphalan IV over 20 minutes on days -4 to -2, antithymocyte globulin (ATG) IV over 4 hours or methylprednisolone IV over 1 hour twice a day on days -3 to -1, and total lymphoid irradiation on day -1. On day 0, patients receive umbilical cord blood (UCB) infusion. Patients with inborn errors of metabolism or inherited hematopoietic disorders receive oral busulfan every 6 hours on days -9 to -6, cyclophosphamide IV over 1 hour on days -5 to -2 or melphalan IV over 20 minutes on days -4 to -2, and ATG IV over 4 hours or methylprednisolone IV over 1 hour on days -3 to -1. On day 0, patients receive UCB infusion. Patients with Fanconi's anemia receive ATG IV over 4 hours or methylprednisolone IV over 1 hour on days -6 to -1, cyclophosphamide IV over 1 hour on days -5 to -2, thoracoabdominal irradiation on day -1, and then the UCB infusion on day 0. Patients also receive cyclosporine and methylprednisolone beginning on day -2 and continuing as necessary as graft-versus-host disease prophylaxis. Patients are followed indefinitely for survival and late toxicity.

PROJECTED ACCRUAL: A total of 4-90 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed diagnosis of one of the following: - Severe aplastic anemia with bone marrow cellularity less than 20% and at least 2 of the following criteria: Granulocyte count less than 500/mm3 Platelet count less than 20,000/mm3 Reticulocyte count less than 50,000/mm3 Etiologies may be Fanconi's anemia, hypoplastic leukemia, monosomy 7, drug exposure (chloramphenicol, NSAIDS), viral exposure (EBV, hepatitis, parvovirus, HIV), nutritional deficiencies, thymoma, paroxysmal nocturnal hemoglobinuria, and amegakaryocytic thrombocytopenia - Myelodysplastic syndrome (MDS) that is refractory to medical management or with cytogenetic abnormalities predictive of transformation into acute leukemia, including 5q-, 7q-, monosomy 7, and trisomy 8 De novo primary or therapy-related secondary MDS Refractory anemia or refractory anemia with ringed sideroblasts only - Inherited hematopoietic disorders that are refractory to medical management Severe combined immunodeficiency Familial erythrophagocytic lymphohistiocytosis Wiskott-Aldrich syndrome Kostmann's syndrome (infantile agranulocytosis) Chronic granulomatous disease Leukocyte adhesion deficiency Chediak-Higashi syndrome Paroxysmal nocturnal hemoglobinuria Fanconi's anemia Dyskeratosis congenita Diamond-Blackfan anemia Amegakaryocytic thrombocytopenia Osteopetrosis Gaucher's disease Lesch-Nyhan syndrome Mucopolysaccharidoses Lipidoses Must also meet all the following conditions: No HLA-ABC/DR identical related bone marrow or UCB donor No 5/6 antigen matched related bone marrow or UCB donor Condition precludes waiting to search and find a donor in the National Marrow Donor Registry Must have backup autologous or haploidentical related marrow Must have available serologic match umbilical cord blood unit in the New York Blood Center's Placental Blood Project

PATIENT CHARACTERISTICS: Age: Not specified Performance status: Zubrod 0-1 OR Karnofsky or Lansky 80-100% Life expectancy: At least 3 months Hematopoietic: See Disease Characteristics Hepatic: Bilirubin no greater than 2.0 mg/dL ALT/AST no greater than 4 times normal Renal: Creatinine no greater than 2.0 mg/dL Creatinine clearance at least 50 mL/min Cardiovascular: Shortening fraction or ejection fraction at least 80% of normal for age Pulmonary: FVC and FEV1 at least 60% predicted for age Adults: DLCO at least 60% predicted Other: No active concurrent malignancy No active infections at time of backup bone marrow harvest or pretransplant cytoreduction Not pregnant or nursing Negative pregnancy test HIV negative

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No concurrent cytotoxic chemotherapy Endocrine therapy: No concurrent immunosuppressive medications Radiotherapy: No concurrent radiotherapy Surgery: Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 1998-08; Primary Completion 2001-01 (Actual); Study Completion 2001-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Jean Bambach, MD, Study Chair — Roswell Park Cancer Institute
Locations (15):
- United States (15):
  - University of Florida Health Science Center, Gainesville, Florida
  - Division of Pediatric Surgery, Jacksonville, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York Blood Center, New York, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of South Carolina School of Medicine, Columbia, South Carolina